CLINICAL TRIAL: NCT02299388
Title: To Evaluate the Effect of Liraglutide on Ambulatory Blood Pressure-A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 523963-1
Record Dates: First submitted 2014-02-04; First posted 2014-11-24 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent; Hypertensive Disease
Keywords: Type 2 Diabetes Mellitus; Hypertension; ambulatory blood pressure monitoring; Endothelial Dysfunction; Pulse pressure; Renin-angiotensin system; heart rate variability
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Active Comparator): All subjects will be advised a low sodium diet. This will be a placebo controlled, double blind and randomized trial of effects of Liraglutide on systolic BP control. Eligible patients will have ABPM measurements and laboratory blood collection at baseline (prior to initiation of Liraglutide or Placebo), at 4 and 8 weeks of therapy. Patients will return 24 hours following ABPM placement for device and data retrieval. Each subject will be asked to keep a log of activities throughout the day.
  Interventions: Drug: Liraglutide or Placebo
- Placebo (Placebo Comparator): All subjects will be advised a low sodium diet. This will be a placebo controlled, double blind and randomized trial of effects of Liraglutide on systolic BP control. Eligible patients will have ABPM measurements and laboratory blood collection at baseline (prior to initiation of Liraglutide or Placebo), at 4 and 8 weeks of therapy. Patients will return 24 hours following ABPM placement for device and data retrieval. Each subject will be asked to keep a log of activities throughout the day.
  Interventions: Drug: Liraglutide or Placebo

INTERVENTIONS:
Drug: Liraglutide or Placebo — All subjects will be advised a low sodium diet. Eligible patients will have ABPM measurements and laboratory blood collection at baseline (prior to initiation of Liraglutide or Placebo), at 4 and 8 weeks of therapy. Patients will return 24 hours following ABPM placement for device and data retrieval.
  Other Names: Victoza

SUMMARY:
The investigators are conducting this research to study the effect of Liraglutide on blood pressure. Several studies have shown increased cardiovascular complications and deaths in diabetics with hypertension. The importance of blood pressure control in diabetes has been shown in many clinical trials. No drug already approved for treating Type 2 Diabetes Mellitus is known to reduce blood pressure along with improving diabetes. However, prior research studies with liraglutide have suggested that treatment with liraglutide improves blood pressure. This effect is seen very quickly and even prior to any weight loss. The mechanism behind this effect is yet to be determined.

DETAILED DESCRIPTION:
The investigators are conducting this research to study the effect of Liraglutide on blood pressure. Several studies have shown increased cardiovascular complications and deaths in diabetics with hypertension. The importance of blood pressure control in diabetes has been shown in many clinical trials. No drug already approved for treating Type 2 Diabetes Mellitus is known to reduce blood pressure along with improving diabetes. However, prior research studies with liraglutide have suggested that treatment with liraglutide improves blood pressure. This effect is seen very quickly and even prior to any weight loss. The mechanism behind this effect is yet to be determined.

Blood pressure will be monitored using the 24 hour Ambulatory Blood Pressure monitor: a device that monitors your blood pressure while you continue normal activity. We have chosen this method to monitor blood pressure because most of the prior studies have proven it to be superior over a single blood pressure recording and its ability to better predict clinical outcomes.

It is well known that both diabetes and hypertension cause endothelial dysfunction. Endothelium is the inner lining of the blood vessels. When it is functioning, it is supposed to regulate blood clotting, help with the body's immune response, controls the volume of fluid and other substances that pass through the blood vessels. Hence, normal endothelial function protects the blood vessels from atherosclerosis (hardening) and builds up of plaque. When it is not functioning well (as in diabetes, hypertension, cigarette smokers etc.) it does not perform one or more of these functions. Hence, in this study, we will also measure the endothelial function using a machine: ENDO PAT.

This is a non-invasive diagnostic test which is done in the doctor's office. Usually takes about 15 minutes. It is not painful. It generates an EndoScore which indicates the current state of the endothelial health.

This is a PILOT study (a small-scale study designed to determine if a larger, full-scale study is doable) to prove this effect which if proven will be extended to a larger, multicenter trial.

Of note: Liraglutide has already been approved for treating Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, as an adjunct to diet and exercise to improve glycemic control (as per approved label.
* HbA1c>7% and ≤10.5% at randomization.
* Men and women of 18-75 years of age.
* Women of childbearing potential must agree to use contraception or must not otherwise be at risk of becoming pregnant. A urine pregnancy test will be done at the time of screening and then every 4 weeks for the duration of 8 weeks. If positive, this will be confirmed with a serum pregnancy test which if positive, appropriate action will be taken as outlined in the detailed protocol.
* Blood pressure≥ 130/80 mm Hg and ≤160/100mmHg on stable treatment (no change in anti hypertensive treatment for 3 months prior to screening) or no treatment. No change in treatment for BP over 8 weeks of the study will be allowed.
* Patient understands the study procedures, alternative treatments are available, and the risks involved with the study, and voluntarily agree to participate by providing written informed consent.

Exclusion Criteria:

* 1. Type 1 diabetes and/or history of ketoacidosis determined by medical history.

  2. History of severe diabetic or autonomic neuropathy, gastroparesis or limb ulceration or amputation.

  3. Therapy with DPP-4 inhibitor, or GLP -1 analog or receptor agonist in the past 6 months.

  4. Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures.

  5. Patients on corticosteroids within 3 months or recurrent continuous corticosteroid treatment (>2 weeks).

  6. Use of weight loss drugs within 3 months of screening or weight loss of ≥10 % in the last 6 months.

  7. Surgery in the past 30 days prior to screening and/or any serious or chronic illness within 6 months or anticipated surgery during the trial period.

  8. Serum creatinine >1.4mg/dL (women)/>1.5mg/dL (men). 9. Serum Triglyceride Level >500 mg/dL. 10. History of pancreatitis. 11. History of drug or alcohol abuse. 12. Poor mental function or any reason to expect patient difficulty in complying with study requirements.

  13. Contraindications to Liraglutide: Personal or family history of medullary thyroid cancer or MEN-2 syndrome 14. Known or suspected allergy to Liraglutide. 15. Diagnosed Secondary hypertension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-10; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Thethi, MD, Principal Investigator — AdventHealth
Locations (1):
- Tulane University Health Science Center, Tidewater building and Tulane Hospital and Clinics, New Orleans, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liraglutide | Placebo
Started | 6 | 5
Completed | 6 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 57.67 [43 to 68] | 59.8 [54 to 66] | 58.64 [43 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 3 | 0 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitors.
Description: To determine whether Liraglutide lowers systolic BP through the day compared to placebo in patients with T2DM who are not on any anti-hypertensive medications or whose BP medications are unchanged over the study period of 8 weeks.
Time Frame: Baseline and 8 Weeks
Population: Only 2 subjects in the placebo group completed 80% ambulatory blood pressure measurements at visits 2 (baseline) and visit 5 (8 weeks).
Measure: Mean (Full Range); unit: mm/Hg
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 6 | 2
mm/Hg | -4.88 [-18.6 to 13.6] | -5.45 [-6.9 to -4.0]

2. Secondary Outcome: Change in Pulse Pressure, Mean Arterial, Diastolic and Nocturnal Blood Pressures.
Description: 1. Change in mean arterial blood pressure and diastolic blood pressure from baseline to 8 weeks in the intent-to-treat (ITT) population.
  2. Change in nocturnal BP: the absence of the nocturnal (between 23:00-06:00 hrs) decline in BP of >/= 10% (defined as "non-dippers") and whether restoration occurs following Liraglutide therapy.
  3. Change in pulse pressure: defined as the difference in systolic and diastolic BPs from baseline to week 8.
Time Frame: Baseline and 8 Weeks
Population: Only 2 subjects in the placebo group completed 80% ambulatory blood pressure measurements at visits 2 (baseline) and visit 5 (8 weeks). One placebo subject did not have an overall pulse pressure value at week 8 and was eliminated from that outcome analysis.
Measure: Mean (Full Range); unit: mm/Hg
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 6 | 2
mm/Hg
  Overall Systolic Pressure | -4.4 [-18.5 to 11.8] | -5.4 [-9.4 to -1.4]
  Overall Diastolic Pressure | -1.8 [-7.5 to 9.5] | -3.3 [-9.8 to 3.2]
  Overall Pulse Pressure: number analyzed (Participants) | 6 | 1
  Overall Pulse Pressure | -2.7 [-11 to 1.4] | 0.4 [0.4 to 0.4]
  Mean Arterial Pressure | -2.6 [-11.2 to 10.3] | -4 [-9.7 to 1.7]
  Nocturnal Systolic Pressure | 1.15 [-18.5 to 14.7] | -2.3 [-25.3 to 20.6]
  Nocturnal Diastolic Pressure | 1.0 [-12.1 to 19] | -0.8 [-14 to 12.5]

3. Other Pre Specified Outcome: Change in Endothelial Function. (Using Endo PAT)
Description: To understand the BP lowering effect of Liraglutide, the investigators will study the Endothelial function - using Endo PAT
Time Frame: Baseline and 8 Weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Autonomic Function (Heart Rate Variability Using Endo PAT.)
Description: To understand the BP lowering effect of Liraglutide, the investigators will study the the autonomic function by assessing the heart rate variability using Endo PAT.
Time Frame: Baseline and 8 Weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Renin-Angiotensin System (Plasma Renin and Aldosterone Levels and Urine Angiotensinogen Levels)
Description: To understand the mechanisms of BP lowering effect of Liraglutide, the investigators will study the effects on Renin Angiotensin system by measuring Plasma renin and aldosterone levels and Urine Angiotensinogen levels (U-AGT-using an assay developed at Tulane Hypertension Center).
Time Frame: Baseline and 8 Weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Catecholamines (Collecting 24 Hrs Urine for Metanephrines and Catecholamines.)
Description: To understand the BP lowering effect of Liraglutide, the investigators will analyse the catecholamines by collecting 24 hrs urine for metanephrines and catecholamines.
Time Frame: Baseline and 8 Weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Urinary Sodium Excretion
Description: To understand the BP lowering effect of Liraglutide, the investigators will assess urinary sodium excretion by collecting 24 hours Urine Sodium.
Time Frame: Baseline and 8 Weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Liraglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No